CLINICAL TRIAL: NCT00258401
Title: The Effectiveness of a Low-Residue Diet on Diarrhea in Cancer Patients Receiving Pelvic Radiation Therapy
Brief Title: Low-Residue Diet in Treating Diarrhea in Patients Receiving Pelvic Radiation Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Amy LeJeune, MS,RD, Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CASE2Z05
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Cervical Cancer; Diarrhea; Prostate Cancer; Radiation Toxicity; Sarcoma
Keywords: diarrhea; radiation toxicity; recurrent uterine sarcoma; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent cervical cancer; stage 0 cervical cancer; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Diarrhea; Prostatic Neoplasms; Radiation Injuries; Sarcoma; Uterine Cervical Dysplasia | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-residue diet (Active Comparator): At the onset of diarrhea symptoms, patients are instructed to eat a low-residue diet. Patients continue on this diet for 2-4 weeks.Patients are interviewed weekly for up to six weeks.
  Interventions: Dietary Supplement: dietary intervention; Procedure: management of therapy complications; Procedure: quality-of-life assessment
- no dietary intervention (Active Comparator): At the onset of diarrhea symptoms, patients undergo no dietary intervention but are interviewed weekly for up to six weeks.
  Interventions: Procedure: management of therapy complications; Procedure: quality-of-life assessment

INTERVENTIONS:
Dietary Supplement: dietary intervention — At the onset of diarrhea symptoms, patients are instructed to eat a low-residue diet. Patients continue on this diet for 2-4 weeks.
  Arms: low-residue diet
Procedure: management of therapy complications — Interviewed weekly for up to 6 weeks to monitor dietary intake, bowel symptoms, diarrhea events, FI-QOL, and changes in CTC scores.
Procedure: quality-of-life assessment — Interviewed weekly for up to 6 weeks to monitor dietary intake, bowel symptoms, diarrhea events, FI-QOL, and changes in CTC scores.

SUMMARY:
RATIONALE: Eating a diet low in residue (fiber, fat, and certain milk or vegetable products) may help prevent or reduce diarrhea caused by pelvic radiation therapy.

PURPOSE: This randomized clinical trial is studying a low-residue diet to see how well it works compared to no dietary intervention in treating diarrhea in patients who are undergoing radiation therapy to the pelvis for uterine, cervical, or prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the nutritional status, Common Toxicity Criteria (CTC) score, and fecal incontinence quality of life (FI-QOL) in patients with uterine, cervical, or prostate cancer who are undergoing pelvic radiotherapy receiving a low-residue diet vs no dietary intervention.
* Compare changes in the CTC score and FI-QOL in patients receiving a low-residue diet vs no dietary intervention.
* Compare the efficacy, in terms of a lower CTC score or higher perceived FI-QOL, of a low-residue diet vs no dietary intervention in these patients.

OUTLINE: This is a parallel, randomized, controlled, pilot study. Patients are stratified according to cancer type. Patients are randomized to 1 of 2 treatment arms.

All patients are interviewed to obtain a baseline grade of diarrhea (according to NCI's Common Toxicity Criteria [CTC] scale) and dietary history and measure Fecal Incontinence Quality of Life (FI-QOL).

* Arm I (intervention): At the onset of diarrhea symptoms, patients are instructed to eat a low-residue diet. Patients continue on this diet for 2-4 weeks. They are interviewed weekly for up to 6 weeks to monitor dietary intake, bowel symptoms, diarrhea events, FI-QOL, and changes in CTC scores.
* Arm II (control): Patients undergo no dietary intervention but are interviewed as in arm I.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of uterine, cervical, or prostate cancer
* Current patient at the Ireland/Case Comprehensive Cancer Center
* Planning pelvic radiation therapy within the next 4 months

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Gastrointestinal

* No enteric support
* No inflammatory bowel disease

Other

* No other concurrent illness or medical condition that would preclude study compliance
* No history of allergies or dietary intolerances (e.g., lactose intolerance) that would preclude study treatment or interfere with study results

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* Concurrent hormonal therapy allowed (e.g., testosterone suppression)

Radiotherapy

* See Disease Characteristics

Surgery

* No prior colectomy

Other

* No concurrent glutamine, psyllium, or other fiber supplements (e.g., Benefiber^® or Metamucil^®)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-05; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Diarrhea as assessed by Fecal Incontinence Questionnaire and CTC v3.0 at baseline and once a week for 6 weeks | baseline and once a week for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amy LeJeune, MS, RD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States